CLINICAL TRIAL: NCT02961127
Title: Association Study to Evaluate TFPI Gene in CAD in Han Chinese
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Yundai Chen, Director of Department of Cardiology, Chinese PLA General Hospital
Other Study IDs: 2013-2-5
Record Dates: First submitted 2016-11-06; First posted 2016-11-10 (Estimated); Last update posted 2016-11-10 (Estimated); Status verified 2016-11

CONDITIONS: Coronary Heart Disease
Keywords: tissue factor pathway inhibitor
MeSH Terms: conditions — Coronary Disease

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Venous blood was collected by standard vein puncture in fasting condition. Four single-nucleotide polymorphisms (SNPs) (rs7586970, rs6434222, rs10153820 and rs8176528) were detected with polymerase chain reaction-direct sequencing method. And the genotypes of these SNPs were determined in both CAD patients and non-CAD controls.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- group 1: no drugs were used in our study
  Interventions: Other: Venous blood was collected
- group 2
  Interventions: Other: Venous blood was collected

INTERVENTIONS:
Other: Venous blood was collected — Venous blood was collected by standard vein puncture in fasting condition

SUMMARY:
The cases were hospitalized patients from two medical centers in Beijing and Harbin respectively. Venous blood was collected by standard vein puncture in fasting condition.

DETAILED DESCRIPTION:
In our study, the CAD was defined by one of the following criteria: (1) based on World Health Organization criteria in terms of elevations of cardiac enzymes, electrocardiography (ECG) and clinical symptoms (angina, chest pressure, or shortness of breath); (2) angiographic evidence of more than 50% stenosis in one or more major coronary arteries; (3) previous history of PCI (percutaneous coronary intervention) or CABG (coronary artery bypass graft). The controls were selected from the two medical centers meeting the following criteria: (1) with no family history for CAD; (2) no clinical symptoms for CAD; (3) resting ECG showed normal results. The subjects with two or more risk factors of CAD (age>45 for man and >55 for woman, hypertension, diabetes, overweight, hyperlipidemia) were subjected to treadmill stress test and selected as controls if their ECG were normal without clinical symptoms. Those with history of cardiomyopathy, valvular disease, peripheral vascular disease, stroke, severe hepatic and kidney deficiency were excluded in our study.

Venous blood was collected by standard vein puncture in fasting condition. Four single-nucleotide polymorphisms (SNPs) (rs7586970, rs6434222, rs10153820 and rs8176528) were detected with polymerase chain reaction-direct sequencing method. And the genotypes of these SNPs were determined in both CAD patients and non-CAD controls.

ELIGIBILITY:
Inclusion Criteria:

The coronary artery disease was defined by one of the following criteria-(1) based on World Health Organization criteria in terms of elevations of cardiac enzymes, electrocardiography (ECG) and clinical symptoms (angina, chest pressure, or shortness of breath); (2) angiographic evidence of more than 50% stenosis in one or more major coronary arteries; (3) previous history of PCI (percutaneous coronary intervention) or CABG (coronary artery bypass graft).

The controls were selected from the two medical centers meeting the following criteria: (1) with no family history for CAD; (2) no clinical symptoms for CAD; (3) resting ECG showed normal results. The subjects with two or more risk factors of CAD (age>45 for man and >55 for woman, hypertension, diabetes, overweight, hyperlipidemia) were subjected to treadmill stress test and selected as controls if their ECG were normal without clinical symptoms.

Exclusion Criteria:

* Those with history of cardiomyopathy, valvular disease, peripheral vascular disease, stroke, severe hepatic and kidney deficiency were excluded in our study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The cases were all hospitalized patients recruited from two medical centers in Beijing and Harbin.
  The participants with two or more risk factors of CAD (age>45 for man and >55 for woman, hypertension, diabetes, overweight, hyperlipidemia) were subjected to treadmill stress test and selected as controls if their ECG were normal without clinical symptoms.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2016-11; Primary Completion 2017-04 (Estimated); Study Completion 2017-05 (Estimated)

PRIMARY OUTCOMES:
the frequencies of TFPI were associated with CAD in Han Chinese | 1 year
  Four single-nucleotide polymorphisms (SNPs) (rs7586970, rs6434222, rs10153820 and rs8176528) were detected with polymerase chain reaction-direct sequencing methods.And the genotypes of these SNPs were determined in both CAD patients and non-CAD controls.

CONTACTS AND LOCATIONS:
Overall Officials: Yundai Chen, Ph D, Study Director — Chinese PLA General Hospital

IPD SHARING:
Plan to Share IPD: No